CLINICAL TRIAL: NCT05627141
Title: Comparison Between Photobiomodulation, Cryotherapy Combined With Compression, and Massage for Muscle Recovery in Crossfit Athletes
Brief Title: Photobiomodulation, Cryotherapy Combined With Compression, and Massage for Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Anhanguera (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Filipe Abdalla dos Reis, PhD, Universidade Anhanguera, Universidade Anhanguera
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2022-03-02; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Laser; Muscle; Fatigue, Heart; Muscle Damage
Keywords: Photobiomodulation; Crossfit; Muscle Damage
MeSH Terms: conditions — Fatigue | interventions — Low-Level Light Therapy; Cryotherapy; Massage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Photobiomodulation (Experimental): 10 participants will receive active photobiomodulation immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage
- Sham Photobiomodulation (Sham Comparator): 10 participants will receive sham photobiomodulation immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage
- Active Cryotherapy (Experimental): 10 participants will receive effective cryotherapy (10-12°C for 20 min) combined with high compression on the lower limbs, or sham (25°C for 20 min) damage and fatigue induction protocol. muscle.
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage
- Sham Cryotherapy (Sham Comparator): 10 participants will receive sham cryotherapy (25°C for 20 min) combined with light compression on the lower limbs immediately after the damage and fatigue induction protocol. muscle.
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage
- Massage (Experimental): 10 participants will receive the effective massage immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session.
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage
- Sham Massage (Sham Comparator): 10 participants will receive the sham massage immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session.
  Interventions: Other: Photobiomodulation; Cryotherapy, Massage

INTERVENTIONS:
Other: Photobiomodulation; Cryotherapy, Massage — Photobiomodulation: the 20 participants will receive active photobiomodulation or sham immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session. Cryotherapy combined with compression: the 20 participants will receive effective cryotherapy (10-12°C for 20 min) combined with high compression, or sham (25°C for 20 min) combined with light compression, on the lower limbs, immediately after the protocol. induction of muscle damage and fatigue. Effective cryotherapy or sham will be applied in a randomized and crossover manner, with an interval of 15 days between each evaluation session.
  Massage: the 20 participants will receive the effective massage or sham immediately after the muscle damage and fatigue induction protocol in a randomized and crossover manner, with an interval of 15 days between each evaluation session.

SUMMARY:
Skeletal muscle fatigue is an inevitable phenomenon in the training and competition routine for many crossfit athletes, which can impair their physical performance and predispose them to musculoskeletal injuries. Thus, strategies and/or therapies that minimize fatigue and accelerate muscle recovery are extremely relevant for everyone involved with sport. The aim of the present study is to investigate and compare the effects of photobiomodulation, cryotherapy combined with compression, and massage as isolated therapies for muscle recovery after a protocol of induced muscle damage and fatigue in Crossfit athletes. This is a randomized, double-blind, crossover, sham-controlled clinical trial. Will be recruited 60 male participants, adults, aged between 18 and 40 years, Crossfit practitioners. They will be randomly allocated into 3 groups of 20 participants per therapy, each crossed between effective and sham every 15 days. The primary outcome will be muscle performance in functional test (free squat) and knee extensor torque in maximal voluntary isometric contraction (MVIC). Secondary outcomes will be evaluated by the levels of muscle damage via creatine phosphokinase (CPK) and inflammatory process via blood C-reactive protein (CRP); and delayed onset muscle pain via numerical verbal scale (0-10). All outcomes will be evaluated at baseline, 24h and 48h after induction of muscle damage and fatigue. Data will be analyzed and compared intra and inter groups with a significance level of 5%.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover, controlled clinical trial of sham therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male participants;
* Adults; aged between 18 and 40 years;
* Body mass index (BMI) between 18 and 30 kg/m2;
* Crossfit practitioners of the scale, amateur, RX and elite categories;
* Training at least 5 days a week.

Exclusion Criteria:

* Orthopedic injuries in the lower limbs (2 months) or during the development of the study will be excluded;
* Participants with less than 5 training sessions per week;
* Participants making regular use of pharmacological agents and/or ergogenic supplements;
* Participants who regularly use alcohol and/or tobacco;
* Participants with skin lesions (open wounds) on the lower limbs.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Force Dynamometry | 48 hours
  participants will be evaluated regarding the dominant knee extensor torque during maximal voluntary isometric contraction (MVIC) in an extensor chair.
Blood markers of muscle damage and inflammatory process | 48 hours
  To measure the serum levels of CPK and CRP, blood samples will be collected after aseptic cleaning of the ventral side of the dominant arm. All blood collection procedures will be performed by a qualified nurse (who will not know to which group each participant will belong). Collections will be performed using vacuum collection tubes, without anticoagulant (10ml), centrifuged at 4,000g for 5 minutes, and stored at -80°C until analysis. Blood collections will be performed at baseline (before WOD and leg extension exercise), 24h and 48h after. Blood analysis will be performed using infrared spectrophotometry in a clinical analysis laboratory (Matter Diagnósticos, Campo Grande, MS) and by an evaluator who is blinded to the therapies applied.
Delayed onset muscle pain | 48 hours
  The subjective perception of pain will be through a numerical verbal scale (NVS) graduated in centimeters (from 0 to 10), where 0 corresponds to no pain, and 10 corresponds to the maximum possible pain (HAWKER et al., 2011). Pain will be provoked in participants through CIVM for knee extension of the dominant lower limb, in full extension (0°) and without load (FERRARESI et al., 2016). Volunteers will be asked about the level of pain they will feel immediately before WOD and MVIC in a leg extension, 24h and 48h after.

CONTACTS AND LOCATIONS:
Overall Officials: Filipe A dos Reis, PhD, Principal Investigator — Ufscar
Locations (1):
- Filipe Abdalla, Campo Grande, Mato Grosso do Sul, Brazil